CLINICAL TRIAL: NCT03702075
Title: Effects of a Self-administered Program in Chronic Neck Pain Patients
Brief Title: Self-administered Program in Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0080UG
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients allocated to the experimental group were included in a self-administered program combining self-myofascial release using foam rollers and roller balls and active upper limb neurodynamic exercises. It consisted of three sessions of 50-60 minutes per week for 4 consecutive weeks.
  Interventions: Other: self-administered program
- Control group (No Intervention): Those patients allocated to the control group received a booklet with information regarding neck pain and explaining basic exercises for active mobilization and stretching with pictures and a short text.

INTERVENTIONS:
Other: self-administered program — One session was a session supervised by a physical therapist in the Faculty of Health Sciences. This session took place in groups of three or four people. All participants had to follow the physiotherapist instructions about the correct way to do the exercises with the foam roller or ball and nerve mobilizations of upper limbs.The other two weekly sessions were performed at home, following the instructions given by the physiotherapist in session.
  Arms: Experimental group

SUMMARY:
Neck pain is a complex biopsychosocial disorder often precipitated or aggravated by neck movements or sustained neck postures. The onset and course of this pain are influenced by environmental and personal factors. Many studies report that participants preferred self-care measures for the management of neck pain and they sought professional help only when those measures fail.

DETAILED DESCRIPTION:
Neck pain is the fourth leading cause of disability worldwide causing an enormous impact on individuals and their families, communities and healthcare systems.While neck pain can be severely disabling and costly, treatment options have shown moderate evidence of effectiveness. No previous study has used foam roller in patients with neck pain. In addition, it has been suggested that neurodynamic interventions provide a peripheral stimulus, reducing the pressure existing within the nerve, improving blood flow, axonal transport and nerve conduction. It was hypothesized that a self-administered intervention focused on myofascial release of main muscles related to neck pain and upper-limb active neurodynamics could reduce the presence of active trigger points and pain, improving functionality and active mobility.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (at least 3 months' duration) not related to trauma of at least 3 on a visual analogue scale
* Participants' symptoms had to be reproduced by median nerve upper-limb neurodynamic test.

Exclusion Criteria:

* Exclusion Criteria:
* Whiplash related neck pain
* Previous cervical surgical intervention
* Cognitive impairments which prevent them to follow instructions
* Visual or acoustic limitations
* Physical therapy in the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Trigger points examination | Change from baseline trigger points examination at 4 weeks
  Trigger points will be explored bilaterally by a blinded assessor in suboccipital, scalene, levator scapulae and upper trapezius muscles

SECONDARY OUTCOMES:
Pain severity | Change from baseline pain at 4 weeks
  Pain will be assessed using the Brief Pain Inventory. It measures the degree of interference of pain with various aspects of life, including mobility and social activities (reactive pain) and pain severity (sensory pain).
Functionality | Change from baseline functionality at 4 weeks
  Functionality will be assessed by the Neck Outcome Score. This is a reliable, valid and responsive measure of self-reported disability for patients with neck pain. It includes 34 items divided into 5 subscales: Mobility, symptoms, sleep disturbance, every day activity and pain and participation in everyday life.
Cervical range of motion | Change from baseline cervical range of motion at 4 weeks
  Cervical range of motion will be measured using a cervical goniometer. Subjects perform neck movements to the fullest extent of their mobility of flexion, extension, right and left lateroflexion, and right and left rotation.
Health related quality of life | Change from baseline health related quality of life at 4 weeks
  Health related quality of life will be measured by euroQol-5D. It contains two sections, a descriptive section and a valuation section.
Fear avoidance beliefs | Change from baseline fear avoidance beliefs at 4 weeks
  Fear avoidance beliefs will be assessed by the the Fear Avoidance Beliefs Questionnaire (FABQ). It consists of 16 sentences related to physical activity (first 5 items) and work (last 11 items).
Anxiety and depression | Change from baseline anxiety and depression at 4 weeks
  Anxiety and depression was evaluated by the the Hospital Anxiety and Depression Scale (HAD).It contains 14 items describing symptoms of depression (7 items) and anxiety (7 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain